CLINICAL TRIAL: NCT03863496
Title: Efficacy of Surgical Treatment by Different Pedicle Screw Systems in Pediatric Neuromuscular Spinal Deformity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ilizarov Center (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ilizarov
Record Dates: First submitted 2019-02-06; First posted 2019-03-05 (Actual); Results first posted 2021-06-10 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-05

CONDITIONS: Neuromuscular Diseases; Neuromuscular Scoliosis
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neuromuscular scoliosis (Other): Efficacy of Surgical Treatment by Different Pedicle Screw Systems in Pediatric Neuromuscular Spinal Deformity
  Interventions: Procedure: Scoliosis surgery

INTERVENTIONS:
Procedure: Scoliosis surgery — All patients will be implanted Medtronic CD Horizon Legacy 4.5 and 5.5 under X-ray control (C-arm), intraoperative spinal deformity surgery safety control and standard anesthetic support.

SUMMARY:
This study was sponsored by Federal state budgetary institution "Russian scientific center for traumatology and orthopedics" n.a. acad. G.A. Ilizarov" of the Ministry of Health of Russian Federation. The study will take place at this center.

It is expected to enroll 70 patients aged 6-25 years with NMD, all of whom will be subjected to thoracic and lumbar spinal deformity surgery.

Patients will be divided into two groups depending on skeletal maturity. The degree of skeletal maturity will be determined on the basis of an X-ray study of spinal and pelvic bones. The type of surgical correction will depend on the group.

DETAILED DESCRIPTION:
First group of patients: local dorsal access. Cranial access: at the level of posterior Th2 5 structures and caudally at the level of L4-S2 vertebrae with exposure of posterior upper spines of iliac wings. Skeletization of vertebrae will be done within transverse processes. Pedicle support points are set bilaterally cranially at each segment level for the space of 3 segments. Caudal support base is formed with pedicle screws in lateral masses of the sacral bone or iliac crests at the level of L5-S1 vertebrae. Control fluorography is performed in two standard planes in order to control screw position. Two "dynamic" rods are formed on the basis of the distance between screw heads allowing 2 cm for distraction; these are two rods connected with a longitudinal connector and bent following the normal sagittal spine profile. After that, channels are formed on both sides under m. erector spinae in the cranial/caudal direction. Pre-bent rods with connectors are placed into the prepared channels. The metal construct is stabilized with internal set screws. If necessary, the construct may be stiffened with crosslinks. Control fluorography is performed in two standard planes in order to control implant position and evaluate correction. The intervention completes with local dorsal spinal fusion with an autobone at the level of base screws. The wound is sewn up in layers tightly.

Group two: dorsal access to the posterior column is gained in accordance with the preoperative plan. The access length depends on the instrumentation area. Vertebral skeletization is performed within transverse processes. Subgroup 1 - pedicle support points are set bilaterally at each segment level. Subgroup 2 - pedicle support points are set bilaterally in every second segment. Segmented instrumentation of 3 cranial segments to prevent dislocation of metal construct elements at the level of Th2-4 or Th3-5 vertebrae is a special measure. Similar to group I, caudal support base is formed with pedicle screws in lateral masses of the sacral bone or iliac crests at the level of L5-S1 vertebrae. Control fluorography is performed after that in two standard planes in order to control screw position. Segmented facetectomy is recommended for additional spine mobilization. Pre-bent rods are placed into support points. Deformity correction is performed by means of a translational maneuver, segmented distraction (concave side) and compression (convex side). The metal construct is stabilized with internal set screws. If necessary, the construct may be stiffened with crosslinks. Control fluorography is performed in two standard planes in order to control implant position and evaluate correction. The intervention completes with dorsal spinal fusion with an autobone along the implants. The postoperative bed is subjected to Redon drain. The drainage is exteriorized to the skin via a separate puncture. The wound is sewn up in layers tightly.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent for participation in the study (separate informed consents for child and parents/caregivers), obtained before conducting any study procedures
* Verified and documented diagnosis (neuromuscular desease, NMD) with the results of neurologic examination
* Deformity of thoracic and/or lumbar spine associated with NMD, which requires surgical intervention

Exclusion Criteria:

* Patient unwillingness or inability to follow study procedures
* Absence of signed and dated informed consent for participation in the study (as for child and for parents/caregivers)
* Patient participation in another clinical study, which can influence the results of this study
* Life expectancy <12 months
* Concomitant diseases, which preclude patient participation in this study according to doctor's opinion

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2021-02-14 (Actual); Study Completion 2021-02-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Ilizarov, Kurgan, Russia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neuromuscular Scoliosis
Started | 71
Completed | 71
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients aged 6 to 22 years with neuromuscular scoliosis
Groups:
- Neuromuscular Scoliosis: Scoliosis surgery: All patients will be implanted with telescopic connector Medtronic CD Horizon Legacy 4.5 and 5.5 under X-ray control (C-arm), intraoperative spinal deformity surgery safety control (NIM Eclipse, Stealth Station S7) and standard anesthetic support.
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 65
  Between 18 and 65 years | 6
  >=65 years | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 14 (3.605)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 45
Race/Ethnicity, Customized [Number; unit: participants]
  Russia | 71
Region of Enrollment [Count of Participants; unit: Participants]
  Russia | 71
Neuromuscular scoliosis [Count of Participants; unit: Participants] | 71

OUTCOME MEASURES:

1. Primary Outcome: First Scoliotic Curve
Description: First scoliotic curve before surgery in Cobb degrees
Time Frame: before surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 69
degrees | 71.4029 (27.60483)

2. Primary Outcome: Second Scoliotic Curve
Description: Second scoliotic curve before surgery in Cobb degrees
Time Frame: before surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 16
degrees | 44,7125 (23,14289)

3. Primary Outcome: Tilt of the Pelvis Relative to the Horizon
Description: tilt of the pelvis relative to the horizon before surgery in Cobb degrees
Time Frame: before surgery
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Neuromuscular Scoliosis: Scoliosis surgery: All patients will be implanted with telescopic connector Medtronic CD Horizon Legacy 4.5 and 5.5 under X-ray control (C-arm), intraoperative spinal deformity surgery safety control and standard anesthetic support.
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 70
degrees | 14.7729 (10.19554)

4. Primary Outcome: Kyphotic Curve Th5-Th12
Description: Kyphotic curve Th5-Th12 before surgery in Cobb degrees
Time Frame: before surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 70
degrees | 28,7029 (24,33570)

5. Primary Outcome: Lordotic Curve L1-S1
Description: Lordotic curve L1-S1 before surgery in Cobb degrees
Time Frame: before surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 70
degrees | 53,8829 (37,75711)

6. Secondary Outcome: First Scoliosis Curve
Description: First scoliotic curve after surgery in Cobb degrees
Time Frame: 10 days after surgery
Measure: Mean (Standard Deviation); unit: degrees
Groups:
- Neuromuscular Scoliosis: Scoliosis surgery: All patients will be implanted Medtronic CD Horizon Legacy 4.5 and 5.5 under X-ray control (C-arm), intraoperative spinal deformity surgery safety control (NIM Eclipse, Stealth Station S7) and standard anesthetic support.
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 69
degrees | 31.4667 (19.21541)

7. Secondary Outcome: Second Scoliotic Curve
Description: Second scoliotic curve after surgery in Cobb degrees
Time Frame: 10 days after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 15
degrees | 28,5533 (15,52168)

8. Secondary Outcome: Tilt of the Pelvis Relative to the Horizon
Description: tilt of the pelvis relative to the horizon after surgery in Cobb degrees
Time Frame: 10 days after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 70
degrees | 6.1514 (5.85862)

9. Secondary Outcome: Kyphotic Curve Th5-Th12
Description: Kyphotic curve Th5-Th12 after surgery in Cobb degrees
Time Frame: 10 days after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 70
degrees | 21,7486 (14,12344)

10. Secondary Outcome: Lordotic Curve L1-S1
Description: Lordotic curve L1-S1 after surgery in Cobb degrees
Time Frame: 10 days after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 70
degrees | 49,6700 (19,06499)

11. Post Hoc Outcome: First Scoliotic Curve
Description: First scoliotic curve 12 months after surgery in Cobb degrees
Time Frame: 12 months after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 44
degrees | 31,6614 (19,25580)

12. Post Hoc Outcome: Second Scoliotic Curve
Description: Second scoliotic curve 12 months before surgery in Cobb degrees
Time Frame: 12 months after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 8
degrees | 28,5750 (23,24065)

13. Post Hoc Outcome: Tilt of the Pelvis Relative to the Horizon
Description: tilt of the pelvis relative to the horizon 12 months after surgery in Cobb degrees
Time Frame: 12 months after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 39
degrees | 7,0513 (6,40924)

14. Post Hoc Outcome: Kyphotic Curve Th5-Th12
Description: Kyphotic curve Th5-Th12 12 months after surgery in Cobb degrees
Time Frame: 12 months after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 43
degrees | 22,9581 (15,93596)

15. Post Hoc Outcome: Lordotic Curve L1-S1
Description: Lordotic curve L1-S1 12 months after surgery in Cobb degrees
Time Frame: 12 months after surgery
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Neuromuscular Scoliosis
Number analyzed (Participants) | 42
degrees | 51.7405 (15.08844)

ADVERSE EVENTS:
Time Frame: 1 year after surgery
Description: implant-dependent complications, Cardiac disorders
Arm/Group | Neuromuscular Scoliosis
All-Cause Mortality (participants affected / at risk) | 1/71
Serious Adverse Events (participants affected / at risk) | 1/71
Other Adverse Events (participants affected / at risk) | 0/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neuromuscular Scoliosis (N=71)
12 months after surgery (Cardiac disorders) | 1 (1) — Sudden death syndrome due to cardiomyopathy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT03863496/Prot_SAP_000.pdf